CLINICAL TRIAL: NCT06851546
Title: Efficacy of Selective Laser Trabeculoplasty Targeting Nasal Versus Inferior 180-degree
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Arthur J. Sit, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-008197
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal 180° Selective Laser Trabeculoplasty (SLT) (Experimental): The Nasal 180° Selective Laser Trabeculoplasty (SLT) will be performed on the right eye.
  After 90 days, the Inferior 180° Selective Laser Trabeculoplasty (SLT) will be performed on the right eye.
  Interventions: Procedure: Nasal 180° Selective Laser Trabeculoplasty (SLT); Procedure: Inferior 180° Selective Laser Trabeculoplasty (SLT)
- Inferior 180° Selective Laser Trabeculoplasty (SLT) (Experimental): The Inferior 180° Selective Laser Trabeculoplasty (SLT) will be performed on the right eye.
  After 90 days, the Nasal 180° Selective Laser Trabeculoplasty (SLT) will be performed on the right eye.
  Interventions: Procedure: Nasal 180° Selective Laser Trabeculoplasty (SLT); Procedure: Inferior 180° Selective Laser Trabeculoplasty (SLT)

INTERVENTIONS:
Procedure: Nasal 180° Selective Laser Trabeculoplasty (SLT) — The Nasal 180° Selective Laser Trabeculoplasty (SLT) will be performed on the right eye. As per standard procedure, the laser will initially be set at 0.8 mJ (or 0.4 mJ for heavily pigmented TM). The energy level will then be adjusted in 0.1 mJ increments: increased until micro-bubble formation is observed or decreased if bubbles are noted. The desired endpoint is the production of a few fine 'champagne bubbles' every 2-3 laser spots. Larger gas bubbles and trabecular meshwork blanching will require the operator to titrate the power downwards in 0.1 mJ increments. Prophylactic IOP lowering and anti-inflammatory drops will be left to physician preference.
Procedure: Inferior 180° Selective Laser Trabeculoplasty (SLT) — The Inferior 180° Selective Laser Trabeculoplasty (SLT) will be performed on the right eye. As per standard procedure, the laser will initially be set at 0.8 mJ (or 0.4 mJ for heavily pigmented TM). The energy level will then be adjusted in 0.1 mJ increments: increased until micro-bubble formation is observed or decreased if bubbles are noted. The desired endpoint is the production of a few fine 'champagne bubbles' every 2-3 laser spots. Larger gas bubbles and trabecular meshwork blanching will require the operator to titrate the power downwards in 0.1 mJ increments. Prophylactic IOP lowering and anti-inflammatory drops will be left to physician preference.

SUMMARY:
The purpose of this study to optimize Selective Laser Trabeculoplasty (SLT) application when used in the management of open angle glaucoma (OAG)

DETAILED DESCRIPTION:
The purpose of this research is to determine the most effective method in using Selective Laser Trabeculoplasty (SLT) for lowering intraocular pressure (IOP) in patients with ocular hypertension or open-angle glaucoma. We will investigate the IOP lowering differences between nasal 180° SLT and inferior 180° SLT,. The second stage will assess the effect of repeating SLT in the opposite 180° sector after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Ability to comprehend the study procedures and agreement to proceed with primary SLT treatment
* Diagnosis of primary or secondary open angle glaucoma or glaucoma suspects with ocular hypertension
* Bilateral disease
* Pre-SLT IOP >21 mmHg measured at least twice during patient's lifetime with or without medication
* Open angles with moderate to intense trabecular pigmentation
* Mild to moderate visual field defects (24-2 standard mean deviations better than the Swedish interactive thresholding algorithm standard of 12 dB)
* No adequate IOP control (low treatment compliance, substantial adverse effects with eyedrops, and at least 2 IOP measurements higher than the individualized target IOP)

Exclusion Criteria:

* Unwilling or unable to give consent
* Unable to attend scheduled post-operative visits
* Previous history of either laser treatment or intraocular surgery, except for non-complicated cataract surgery (performed >6 months before SLT)
* History of ocular trauma
* Narrow angles
* Retinal detachment
* Active iris neovascularization or active proliferative retinopathy
* Active uveitis
* Monocular patients
* Current use of steroids (ocular, periocular, or systemic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Difference in mean intraocular pressure (IOP) | Baseline, 3 months, 6 months, 9 months
  During each visit, two consecutive IOP measurements will be obtained per eye, and the average of these values will be reported.

SECONDARY OUTCOMES:
Change in intraocular pressure (IOP) | Baseline, 3 months, 6 months, 9 months
  Change in intraocular pressure (IOP), reported as a percentage
Intraocular pressure (IOP) lowering eye drops | 9 months
  Total number of patients that did not need intraocular pressure (IOP) lowering drops after the selective laser trabeculoplasty (SLT)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Sit, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States
- Eye Care Centre, Victoria General Hospital, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials